CLINICAL TRIAL: NCT04974723
Title: A Retrospective, Observational Cohort Study Evaluating the Effectiveness and Cardiovascular Safety of Abaloparatide in Postmenopausal Women New to Anabolic Therapies
Brief Title: Real-world Effectiveness and Cardiovascular Safety Study of Abaloparatide in Postmenopausal Women
Status: Completed | Type: Observational
Sponsor: Radius Health, Inc. (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: BA058-05-028
Record Dates: First submitted 2021-06-18; First posted 2021-07-23 (Actual); Results first posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2023-10

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — abaloparatide; Teriparatide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients Treated with Abaloparatide: Patients who filled ≥ 1 prescription for ABL (TYMLOS) as their index medication during the identification period.
  Interventions: Drug: Abaloparatide
- Patients Treated with Teriparatide: Patients who filled ≥ 1 prescription for TPTD (Forteo) as their index medication during the identification period.
  Interventions: Drug: Teriparatide

INTERVENTIONS:
Drug: Abaloparatide — Abaloparatide subcutaneous (abaloparatide SC [ABL]; Tymlos®)
  Other Names: Tymlos
  Groups: Patients Treated with Abaloparatide
Drug: Teriparatide — Teriparatide subcutaneous (TPTD; Forteo®)
  Other Names: Forteo
  Groups: Patients Treated with Teriparatide

SUMMARY:
The purpose of the study is to evaluate the real-world effectiveness and cardiovascular safety of ABL compared with TPTD during the 18-month period after treatment initiation in propensity score (PS)-matched cohorts

DETAILED DESCRIPTION:
This is a retrospective observational cohort study using healthcare administrative claims data from the USA.

This study will use anonymized patient claims data from PRA's Symphony Health Patient Source Integrated Dataverse (IDV) database including the enhanced hospital data. Data are routinely collected in healthcare encounters from all available healthcare sites (inpatient hospital, outpatient hospital, physician office, pharmacy, etc.) for all types of provided services including specialty, preventive care, and office-based treatments.

The patients for inclusion in the study analyses will be identified based on the prescribed anabolic therapy filled (ABL or TPTD). The identification period (May 1, 2017 to June 30, 2019) was chosen to coincide with the date of the FDA approval of ABL in the USA.

ELIGIBILITY:
Inclusion Criteria:

* Women who are 50 years or older
* ≥1 prescription fill for ABL or TPTD during the identification period
* ≥ 1 claim for medical or hospital visit and a pharmacy claim in the 12 months before the index date

Exclusion Criteria:

* Paget's disease
* Malignancy, except for nonmelanoma skin cancers, carcinoma in-situ of the cervix, ductal carcinoma in-situ of breast
* Indicators of high disease burden and high risk of death
* With prior index anabolic treatment
* Switch to a different anabolic treatment after index date

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study eligibility criteria are in alignment with the prescribing information in the FDA approved labels for both ABL and TPTD and include women with postmenopausal osteoporosis.
Sampling Method: Probability Sample
Enrollment: 22054 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Radius Health, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cosman F, Cooper C, Wang Y, Mitlak B, Varughese S, Williams SA. Comparative effectiveness and cardiovascular safety of abaloparatide and teriparatide in postmenopausal women new to anabolic therapy: A US administrative claims database study. Osteoporos Int. 2022 Aug;33(8):1703-1714. doi: 10.1007/s00198-022-06413-y. Epub 2022 May 7. PMID 35524068

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Propensity score (PS) matching was used to create treatment cohorts. Patients were matched using an extensive list of indicators of disease severity and fracture risk, including fracture and treatment history, as well as conditions associated with increased risk of fall and the requirement for treatments associated with poor bone health or quality.
Groups:
- Patients Treated With Abaloparatide: Patients who filled ≥ 1 prescription for Abaloparatide (ABL) (TYMLOS) as their index medication during the identification period.
- Patients Treated With Teriparatide: Patients who filled ≥ 1 prescription for Teriparatide (TPTD) (Forteo) as their index medication during the identification period.
Period: Overall Study
Arm/Group | Patients Treated With Abaloparatide | Patients Treated With Teriparatide
Started | 11027 | 11027
Completed (This study is a retrospective claims-based cohort study, patients included in the analyses did not actively participate in the study and no study visits were required.) | 11027 | 11027
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients meeting the study inclusion/exclusion criteria and selected after PS-matching.
Groups:
- Patients Treated With ABL: Patients who filled ≥ 1 prescription for ABL (TYMLOS) as their index medication during the identification period.
- Patients Treated With TPTD: Patients who filled ≥ 1 prescription for TPTD (Forteo) as their index medication during the identification period.
- Total: Total of all reporting groups
Arm/Group | Patients Treated With ABL | Patients Treated With TPTD | Total
Number analyzed (Participants) | 11027 | 11027 | 22054
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (8.35) | 67.4 (8.39) | 67.38 (8.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11027 | 11027 | 22054
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 144 | 150 | 294
  Asian | 100 | 104 | 204
  White | 4137 | 4262 | 8399
  Hispanic | 646 | 531 | 1177
  Other | 127 | 107 | 234
  Unknown | 5873 | 5873 | 11746

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Nonvertebral Fracture
Description: A nonvertebral fracture is any fragility fracture at the hip, pelvis, femur, ankle, shoulder (including shoulder, humerus, clavicle), radius/ulna, wrist, or tibia/fibula. The date of the first prescription claim for either abaloparatide or teriparatide during the identification period was considered the index date. A claims-based algorithm with high specificity for fracture site was used to identify osteoporosis related fractures. Patients were followed for up to 18 months after their index date, plus 30 days follow-up or until their first nonvertebral fracture event or hospital death, whichever came first.
Time Frame: From index date up to 19 months
Population: All patients meeting the study inclusion/exclusion criteria and selected after PS-matching.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Treated With ABL | Patients Treated With TPTD
Number analyzed (Participants) | 11027 | 11027
Participants | 313 | 333
Statistical Analysis 1: Comparison: Patients Treated With ABL vs Patients Treated With TPTD; Test type: Non-Inferiority — Cox proportional hazard model was used to calculate the hazard ratio with teriparatide as reference. Noninferiority of abaloparatide to teriparatide was to be concluded if the upper bound of the 2-sided 95% CI of the HR between abaloparatide versus teriparatide was <1.3; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.81 to 1.10]

2. Secondary Outcome: Number of Participants With Composite Endpoint of Nonfatal Myocardial Infarction (MI), Nonfatal Stroke, or In-hospital Cardiovascular Death
Description: Cardiovascular safety was evaluated based only on events occurring from the beginning of the index period through 19 months. The date of the first prescription claim for either abaloparatide or teriparatide during the identification period was considered the index date. Cardiovascular events (MI and stroke) were defined as the first post-index incidence recorded on a hospital claim or physician claim. A validated claims-based algorithm was used to identify deaths, based on hospital discharge status, that are likely to be caused by cardiovascular events. Patients were followed for up to 18 months while on treatment plus 30 days follow-up, or until their first cardiovascular event (MI or stroke) or hospital death, whichever came first.
Time Frame: From index date up to 19 months
Population: All patients meeting the study inclusion/exclusion criteria and selected after PS-matching.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Treated With ABL | Patients Treated With TPTD
Number analyzed (Participants) | 11027 | 11027
Participants | 221 | 211
Statistical Analysis 1: Comparison: Patients Treated With ABL vs Patients Treated With TPTD; Cox proportional hazard model was used to calculate the hazard ratio with teriparatide as reference. Noninferiority of abaloparatide to teriparatide was to be concluded if the upper bound of the 2-sided 95% CI of the HR between abaloparatide versus teriparatide was <1.3; Test type: Superiority; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.89 to 1.30]

3. Secondary Outcome: Number of Participants With a Composite Endpoint of Nonfatal MI, Nonfatal Stroke, Heart Failure or In-hospital Cardiovascular Death
Description: Cardiovascular safety was evaluated based only on events occurring from the beginning of the index period through 19 months. The date of the first prescription claim for either abaloparatide or teriparatide during the identification period was considered the index date. Cardiovascular events (MI, stroke, and heart failure) were defined as the first post-index incidence recorded on a hospital claim or physician claim. A validated claims-based algorithm was used to identify deaths, based on hospital discharge status, that are likely to be caused by cardiovascular events. Patients were followed for up to 18 months while on treatment plus 30 days follow-up, or until their first cardiovascular event (MI, stroke, or heart failure) or hospital death, whichever came first.
Time Frame: From index date up to 19 months
Population: All patients meeting the study inclusion/exclusion criteria and selected after PS-matching.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Treated With ABL | Patients Treated With TPTD
Number analyzed (Participants) | 11027 | 11027
Participants | 495 | 471
Statistical Analysis 1: Comparison: Patients Treated With ABL vs Patients Treated With TPTD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.95 to 1.22]

4. Other Pre Specified Outcome: Number of Participants With Hip Fracture
Description: The date of the first prescription claim for either abaloparatide or teriparatide during the identification period was considered the index date. A claims-based algorithm with high specificity for fracture site was used to identify osteoporosis related fractures. Patients were followed up for 18 months after their index date, plus 30 days follow-up or until their first hip fracture event or hospital death, whichever came first.
Time Frame: From index date up to 19 months
Population: All patients meeting the study inclusion/exclusion criteria and selected after PS-matching.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Treated With ABL | Patients Treated With TPTD
Number analyzed (Participants) | 11027 | 11027
Participants | 112 | 125

ADVERSE EVENTS:
Time Frame: From index date up to 19 months
Description: The design of this study was characterized by secondary use of data previously collected from health insurance claims. Thus, "Serious Adverse Events" and "Other (Not Including Serious) Adverse Events" data was not collected. Only deaths recorded on the hospital discharge status were available and are presented in the "All-Cause Mortality" section below. Date of the first prescription claim for either abaloparatide or teriparatide during the identification period was considered the index date.
Arm/Group | Patients Treated With ABL | Patients Treated With TPTD
All-Cause Mortality (participants affected / at risk) | 10/11027 | 9/11027
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This was a non-controlled, non-randomized study. The data source was administrative claims data that was not collected for research purposes and included potential inaccuracies related to use of prescription medications. Only deaths recorded on the hospital discharge status were available for the derivation of cardiovascular death in this study. Detailed clinical data such as BMD values were not available, and unknown confounding factors were not adjusted for in propensity score matching.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-09): https://cdn.clinicaltrials.gov/large-docs/23/NCT04974723/Prot_SAP_000.pdf